CLINICAL TRIAL: NCT03291028
Title: Defining the Genomic and Histologic Landscape of Primary and Metastatic Tumors With Divergent Kinetics in Patients With Renal Cell Carcinoma (RCC) and Urothelial Carcinoma (UC) Treated With Immune Checkpoint Blockade (ICB)
Brief Title: Analysis of Primary and Metastatic Tumors in Patients With Renal Cell Carcinoma and Urothelial Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: GU-118
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Renal Cell Carcinoma; Urothelial Carcinoma; Bladder Cancer; Ureter Cancer; Urethral Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsied/ resected tumor samples that have been stored in the biosample repository would be used for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with immune check point blocker: Patients who were treated with immune checkpoint inhibitor targeting PD1 and developed metastatic lesion later
  Interventions: Biological: Immune checkpoint inhibitor targeting PD1
- Patients treated with targeted/ observational therapy: Patients who were not treated with immune checkpoint inhihibitor and developed metastatic lesion following other targeted therapy

INTERVENTIONS:
Biological: Immune checkpoint inhibitor targeting PD1 — RCC and UC patients treated with immune checkpoint blockade
  Groups: Patients treated with immune check point blocker

SUMMARY:
This is a comparative study using resected/ biopsied tumors samples collected from renal cell carcinoma and urothelial carcinoma patients who underwent surgical removal of lesions, followed by immune checkpoint blockade (ICB) treatment targting programmed cell death 1 (PD1) but developed new lesions later were also removed and stored in the biosample repository (BSR). The histology and genomic analysis of the pre-treatment and metastatic samples from the same patient would be used to find out the changes that may have lead to metastasis. Also, metastatic samples from ICB naive patients would be collected and compared with those from ICB treated patients to find out if the metastasis in treated patients was due to development of reistance.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include retrospectively identified patients with RCC or UC who have received treatment with ICB and achieved clinical benefit but subsequently developed a solitary new/progressive lesion that was removed surgically. Patients with other tumor types who otherwise meet criteria may be included at a later time
* Additionally, a group of patients with RCC who have undergone a metastasectomy but who did not receive treatment with ICB will be identified. These patients may be approached for study participation to serve as a comparator group

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RCC and UC patients who were treated with ICB but developed metastatis post-treatment that was resected
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Histopathological characterization of samples from ICB treated patients | 18 months
  To characterize differences in histopathology and patterns of genomic expression between baseline tumors and metastases exhibiting divergent growth kinetics ("escape" metastases) in patients treated with immune checkpoint blockade (ICB)
Genomic characterization of samples from ICB treated patients | 18 months
  To characterize expression of different genes between baseline tumors and metastases exhibiting divergent growth kinetics ("escape" metastases) in patients treated with immune checkpoint blockade (ICB)

SECONDARY OUTCOMES:
Histopathological characterization of samples from patients treated with targeted or observational therapy | 18 months
  To characterize differences in histopathology between baseline tumors and metastases in patients with RCC treated with observation or targeted therapy.
Comparison of Histopathological characteristics of metastatic samples from ICB naive and treated patients | 18 months
  To characterize differences in histopathology and patterns of genomic expression between "escape" metastases in patients treated with ICB from patients treated with targeted therapy or observation.
Genomic characterization of samples from patients treated with targeted or observational therapy | 18 months
  To characterize differences in patterns of genomic expression between baseline tumors and metastases in patients with RCC treated with observation or targeted therapy
Comparison of genomic characteristics of metastatic samples from ICB naive and treated patients | 18 months
  To characterize differences in patterns of genomic expression between "escape" metastases in patients treated with ICB from patients treated with targeted therapy or observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States